CLINICAL TRIAL: NCT05289414
Title: Clinical Efficacy of Pulsed Radiofrequency Treatment Targeting the Mid Cervical Medial Branches Versus Greater Occipital Nerve for Cervicogenic Headache
Brief Title: Pulsed Radiofrquency Targeting Mid Cervical Medial Branches Versus GON for Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HAAbdelhafeez, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PRF GON vs midcervical in CEH
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: two groups of patients diagnosed with cervicogenic headache Will be randomly subjected to either RF on greater occipital nerve or mid cervical medial branches
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple blind study (participant ,investigator and outcome assessor) will be masked and will not konw what is the type of treatment patients receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF on mid cervical medial branches (Active Comparator): first group of patients will be sujected to pulsed radiofrequency on mid cervical medial branches
  Interventions: Device: Radiofrequency on mid cervical medial branches
- PRF on greater occipital nerve (Active Comparator): second group of patients will be subjected to pulsed radiofrequency on Greater occipital nerve
  Interventions: Device: Radiofrequency

INTERVENTIONS:
Device: Radiofrequency on mid cervical medial branches — patients with diagnosis of cervicogenic headache will be subjected to radiofrequency on mid cervical medial branches
  Arms: PRF on mid cervical medial branches
Device: Radiofrequency — patients with diagnosis of cervicogenic headache will be subjected to radiofrequency on Greater occipital nerve
  Arms: PRF on greater occipital nerve

SUMMARY:
To detect the Clinical efficacy of pulsed radiofrequency treatment targeting the mid cervical medial branches versus greater occipital nerve for cervicogenic headache

DETAILED DESCRIPTION:
Cervicogenic headache (CHA) is one of the secondary headache disorders. The prevalence of CHA was estimated to be ~4.1%, and most of the patients affected by CHA report un-resolved, recurrent throbbing pain.

it has been treated with many treatment modalities, such as the administration of medi-cines, physiotherapy, transcutaneous electrical nerve stimulation, and interventional pro-cedures. However, these treatments do not result in long-term relief for many patients and need to be repeated Pulsed radiofrequency treatment (PRF) is one of the modalities used to treat CHA

. CHA has been known to originate from the convergence of the 3 upper cervical and tri-geminal afferents, and therefore, many physicians have performed PRF targeting the upper cervical structures (occipital nerve, C2 dorsal root ganglion).

However, this results in only short-term pain relief in the posterior head, and it can lead to some complications, such as vascular and nerve injuries. Because of these limitations, we will attempt PRF targeting the mid-cervical medial branches

ELIGIBILITY:
Inclusion Criteria:

1. medically stable outpatients with confirmed diagnosis of cervicogenic headache according to International Headache society
2. Are reliable and willing to make themselves available for the duration of the study and are willing to follow up.
3. Men or women older than 18years of age .
4. clear written informed consent from each participant in the trial.

Exclusion Criteria: 1)pregnants, breastfeeding, or willing to be pregnant during the study.

2)presence of clinically significant medical or psychiatric condition that may increase the risk associated with the study 3)participation in any other type of medical research that may interfere with the interpretation of the study.

4)patients with haemocoagulation disorders, local infection or those who refused to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) | 6 months
  Assessment of pain will be done using VAS The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Visual analogue scale | 3 months
visual analogue scale | 1 month
visual analogue scale | 2 weeks
visual analogue scale | 48 hours
patient satisfactory score | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sjaastad O, Bakketeig LS. Prevalence of cervicogenic headache: Vaga study of headache epidemiology. Acta Neurol Scand. 2008 Mar;117(3):173-80. doi: 10.1111/j.1600-0404.2007.00962.x. Epub 2007 Nov 20. PMID 18031563
- [Background] Chua NH, Vissers KC, Sluijter ME. Pulsed radiofrequency treatment in interventional pain management: mechanisms and potential indications-a review. Acta Neurochir (Wien). 2011 Apr;153(4):763-71. doi: 10.1007/s00701-010-0881-5. Epub 2010 Nov 30. PMID 21116663
- [Background] Hamer JF, Purath TA. Response of cervicogenic headaches and occipital neuralgia to radiofrequency ablation of the C2 dorsal root ganglion and/or third occipital nerve. Headache. 2014 Mar;54(3):500-10. doi: 10.1111/head.12295. Epub 2014 Jan 16. PMID 24433241
- [Background] Palea O, Andar HM, Lugo R, Granville M, Jacobson RE. Direct Posterior Bipolar Cervical Facet Radiofrequency Rhizotomy: A Simpler and Safer Approach to Denervate the Facet Capsule. Cureus. 2018 Mar 14;10(3):e2322. doi: 10.7759/cureus.2322. PMID 29765790